CLINICAL TRIAL: NCT00184847
Title: Adenosine Receptor Involvement in Acute Ischemic Preconditioning of the Vascular Endothelium
Brief Title: Adenosine Receptors Influence Ischemia-Reperfusion Injury
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: ACAD
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Ischemia-Reperfusion Injury
Keywords: acetylcholine; adenosine; caffeine; ischemic preconditioning
MeSH Terms: conditions — Reperfusion Injury | interventions — Acetylcholine; Adenosine; Caffeine

INTERVENTIONS:
Drug: acetylcholine
Procedure: twenty minutes of forearm ischemia
Procedure: three 5-minute periods of forearm ischemia
Drug: adenosine
Drug: caffeine

SUMMARY:
Ischemic preconditioning is defined as the development of tolerance to ischemia-reperfusion injury by a previous short bout of ischemia resulting in a marked reduction in infarct size. This mechanism can be mimicked by several pharmacological substances such as acetylcholine and adenosine.

To detect ischemia-reperfusion injury in humans in vivo Kharbanda et al. developed a method in which endothelial dysfunction represents the effects of ischemic preconditioning. This method, however, uses acetylcholine to measure endothelial function before and after forearm ischemia. We, the investigators at Radboud University, hypothesize that the use of acetylcholine in this model reduces ischemia-reperfusion injury. Therefore, we will compare this protocol with a protocol in which endothelial function is only measured after ischemia. We expect an increase in ischemia-reperfusion injury when endothelial function is only measured after the forearm ischemia.

After determining the optimal method to measure ischemia-reperfusion injury of the vascular endothelium we will determine the effect of acute and chronic caffeine, an adenosine receptor antagonist, on ischemic preconditioning. With this study we expect to find that adenosine mimics ischemic preconditioning of the vascular endothelium. Moreover, we expect to find that acute caffeine intake reduces ischemia-reperfusion injury whereas chronic caffeine intake does not. This study will increase our knowledge about the mechanism of ischemic preconditioning and may also provide leads to exploit this endogenous protective mechanism in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2005-03

PRIMARY OUTCOMES:
Percentual increase in forearm blood flow ratio to three increment dosages of acetylcholine before forearm ischemia and within two hours after forearm ischemia

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Rongen, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Centre/Department of Pharmacology and Toxicology
Locations (1):
- Radboud University Nijmegen Medical Centre/Department of Pharmacology and Toxicology, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Kharbanda RK, Peters M, Walton B, Kattenhorn M, Mullen M, Klein N, Vallance P, Deanfield J, MacAllister R. Ischemic preconditioning prevents endothelial injury and systemic neutrophil activation during ischemia-reperfusion in humans in vivo. Circulation. 2001 Mar 27;103(12):1624-30. doi: 10.1161/01.cir.103.12.1624. PMID 11273988